CLINICAL TRIAL: NCT04654468
Title: A Phase III, Multicenter, Single Arm Study Evaluating the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Crovalimab in Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH) Not Previously Treated With Complement Inhibition
Brief Title: A Study Evaluating the Efficacy, Safety, Pharmacokinetics and Pharmacodynamics of Crovalimab in Participants With Paroxysmal Nocturnal Hemoglobinuria (PNH) Not Previously Treated With Complement Inhibition
Acronym: COMMODORE 3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YO42311
Record Dates: First submitted 2020-11-30; First posted 2020-12-04 (Actual); Results first posted 2023-06-05 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Crovalimab (Experimental): Participants will receive a loading series of crovalimab comprised of an intravenous (IV) dose on Day 1, followed by weekly crovalimab subcutaneous (SC) doses for 4 weeks on Week 1 Day 2, then on Weeks 2, 3, and 4. Maintenance SC dosing will begin at Week 5 and will continue Q4W (every 4 weeks) thereafter for a total of 24 weeks of study treatment. After 24 weeks of crovalimab treatment, participants who derive benefit from the drug may continue to receive crovalimab.
  Interventions: Drug: Crovalimab

INTERVENTIONS:
Drug: Crovalimab — Crovalimab will be administered at a dose of 1000 milligrams (mg) IV (for participants with body weight between 40 and 100 kg) or 1500 mg IV (for participants with body weight ≥ 100 kg) on Week 1 Day 1. On Week 1 Day 2 and on Weeks 2, 3 and 4, it will be administered at a dose of 340 mg SC. For Week 5 and Q4W thereafter, it will be administered at a dose of 680 mg SC (for participants with body weight between 40 and 100 kg) or 1020 mg SC (for participants with body weight ≥ 100 kg). Dosing schedule will be as described above.

SUMMARY:
This study will enroll participants aged 12 years or older with a body weight ≥ 40 kilograms (kg) diagnosed with PNH who have not been previously treated with complement inhibitor therapy. Approximately 50 participants will be treated with Crovalimab for at least 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Body weight ≥ 40 kg at screening
* Willingness and ability to comply with all study visits and procedures
* Documented diagnosis of PNH, confirmed by high sensitivity flow cytometry
* LDH Levels ≥ 2x the ULN at screening
* Participants who have at least four transfusions during 12 months prior to screening (documented in the medical record)
* Presence of one or more of the PNH-related signs or symptoms within 3 months of screening
* Vaccination against Neisseria meningitidis serotypes A, C, W, and Y < 3 years prior to initiation of study treatment (Day 1)
* Vaccination against Haemophilius influenzae type B and Streptococcus pneumonia according to national vaccination recommendations
* For participants receiving other therapies (e.g., immunosuppressants, corticosteroids): stable dose for ≥ 28 days prior to screening and up to the first drug administration
* Adequate hepatic and renal function
* Women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception during the treatment period and for 46 weeks (approximately 10.5 months) after the final dose of crovalimab
* Platelet count ≥30,000 per cubic millimeter (mm^3) at screening
* ANC > 500/microlitres (μl) at screening

Exclusion Criteria:

* Current or previous treatment with a complement inhibitor
* History of allogeneic bone marrow transplantation
* History of Neisseria meningitidis infection within 6 months prior to screening and up to first drug administration
* Known or suspected immune or hereditary complement deficiency
* Known HIV infection with cluster of differentiation 4 (CD4) count < 200 cells/µl within 24 weeks prior to screening
* Infection requiring hospitalization or treatment with IV antibiotics within 28 days prior to screening and up to the first drug administration, or oral antibiotics within 14 days prior to screening and up to the first drug administration
* Active systemic bacterial, viral, or fungal infection within 14 days before first drug administration
* Presence of fever (≥ 38˚C) within 7 days before the first drug administration
* Splenectomy < 6 months before screening
* History of malignancy within 5 years prior to screening and up to the first drug administration
* Pregnant or intending to become pregnant during the study or within 46 weeks (10.5 months) after the final dose of study treatment
* Participation in another interventional treatment study with an investigational agent or use of any experimental therapy within 28 days of screening or within 5 half-lives of that investigational product, whichever is greater

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2026-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- China (4):
  - West China Hospital, Sichuan University, Chengdu
  - Institute of Hematology and Hospital of Blood Disease, Tianjin
  - Tianjin Medical University General Hospital, Tianjin
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Roth A, Fu R, He G, Alzahrani H, Chou SC, Hicheri Y, Kazmierczak M, Recova VL, Uchiyama M, Vladareanu AM, Beveridge L, Buatois S, Buri M, Compagno N, Shi D, Balachandran N, Sreckovic S, Scheinberg P. Safety of Crovalimab Versus Eculizumab in Patients With Paroxysmal Nocturnal Haemoglobinuria (PNH): Pooled Results From the Phase 3 COMMODORE Studies. Eur J Haematol. 2025 Feb;114(2):373-382. doi: 10.1111/ejh.14339. Epub 2024 Nov 13. PMID 39535306
- [Derived] Liu H, Xia L, Weng J, Zhang F, He C, Gao S, Jia J, Chang AC, Lundberg P, Shi J, Sima CS, Sostelly A, Sreckovic S, Xiao Z, Zhang Z, Fu R. Efficacy and safety of the C5 inhibitor crovalimab in complement inhibitor-naive patients with PNH (COMMODORE 3): A multicenter, Phase 3, single-arm study. Am J Hematol. 2023 Sep;98(9):1407-1414. doi: 10.1002/ajh.26998. Epub 2023 Jul 8. PMID 37421604

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 5 investigative sites in China.
Pre-assignment Details: A total of 51 participants with a diagnosis of paroxysmal nocturnal hemoglobinuria (PNH) were enrolled in the study and received at least 1 dose of crovalimab.
Groups:
- Crovalimab: Crovalimab was administered at an initial loading dose of 1000 milligrams (mg) (for participants with body weight between 40 and 100 kg) or 1500 mg (for participants with body weight >=100kg), as intravenous (IV) injection on Day 1 of Week 1 followed by four weekly subcutaneous (SC) injections of 340 mg starting on Day 2 of Week 1 and then once weekly (QW) at Weeks 2,3 and 4. Thereafter crovalimab was administered, as SC injection, at a maintenance dose of 680 mg (for participants with body weight between 40 and 100kg) or 1020 mg (for participants with body weight >=100kg) once every 4 weeks (Q4W) from Week 5 for a total of 24 weeks of study treatment. Participants who derive benefit from the drug after 24 weeks of treatment may continue to receive crovalimab Q4W.
Period: Overall Study
Arm/Group | Crovalimab
Started | 51
Completed | 0
Not Completed | 51
Not completed — Death | 1
Not completed — Ongoing in the Study | 50

BASELINE CHARACTERISTICS:
Population: Safety population included all enrolled participants who received at least one dose of crovalimab.
Groups:
- Crovalimab: Crovalimab was administered at an initial loading dose of 1000 mg (for participants with body weight between 40 and 100) kg or 1500 mg (for participants with body weight >=100kg), as IV injection on Day 1 of Week 1 followed by four weekly SC injections of 340 mg starting on Day 2 of Week 1 and then QW at Weeks 2,3 and 4. Thereafter crovalimab was administered, as SC injection, at a maintenance dose of 680 mg (for participants with body weight between 40 and 100kg) or 1020 mg (for participants with body weight >=100kg) Q4W from Week 5 for a total of 24 weeks of study treatment. Participants who derive benefit from the drug after 24 weeks of treatment may continue to receive crovalimab.
Arm/Group | Crovalimab
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.0 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 51
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 51
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Percentage of Participants With Hemolysis Control
Description: A Generalized Estimating Equation (GEE) was used to estimate the population-average percentage of the participants with hemolysis control (measured by lactate dehydrogenase (LDH) ≤1.5 x upper limit of normal (ULN)) from Week 5 to Week 25 taking account of the intra-patient and inter-patient correlation between LDH control statuses across visits. The dependent variable was the binary indicator for hemolysis control. Independent variables are categorical effects of visits, continuous baseline LDH.
Time Frame: From Week 5 up to Week 25
Population: Primary Analysis Population (PAP) included all enrolled participants who received at least one dose of crovalimab and had at least one central LDH level assessment after the first IV infusion.
Measure: Least Squares Mean (95% Confidence Interval); unit: mean percentage of participants
Arm/Group | Crovalimab
Number analyzed (Participants) | 51
mean percentage of participants | 78.66 [67.78 to 86.59]

2. Primary Outcome: Difference in Percentage of Participants With Transfusion Avoidance (TA) From Baseline Through Week 25 and Within 24 Weeks Prior to Screening
Description: TA was defined as participants who were packed red blood cell (pRBC) transfusion-free and did not require transfusion per protocol-specified guidelines. TA within 24 weeks prior to screening was based on the pRBC transfusion history in the medical records. Reported in this outcome measure is the difference in the percentage of participants between "baseline through Week 25" and "within 24 weeks prior to screening". 95% Confidence Interval (CI) for the difference between the percentage of participants with transfusion avoidance between Pre-screening and Post-baseline is calculated using the Newcombe method.
  Screening= Day -28 to Day -1 and Baseline= Day 1.
Time Frame: 24 Weeks Prior to Screening, Baseline to Week 25
Population: PAP included all enrolled participants who received at least one dose of crovalimab and had at least one central LDH level assessment after the first IV infusion.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Crovalimab
Number analyzed (Participants) | 51
percentage of participants | 50.98 [34.30 to 65.05]
Statistical Analysis 1: Comparison: Crovalimab; Percentage of participants who achieved TA from baseline through Week 25 were compared with the percentage of participants who reported TA within 24 weeks prior to screening; Test type: Superiority; p < .0001, Paired McNemar

3. Secondary Outcome: Percentage of Participants With Breakthrough Hemolysis (BTH)
Description: BTH was defined as at least one new or worsening symptom or sign of intravascular hemolysis (fatigue, hemoglobinuria, abdominal pain, shortness of breath [dyspnea], anemia [hemoglobin < 10 grams per deciliter (g/dL)], major adverse vascular event [MAVE, including thrombosis], dysphagia, or erectile dysfunction) in the presence of elevated LDH ≥2xULN after a prior LDH reduction to ≤1.5xULN from the start of study treatment. As pre-specified in the SAP participants withdrawing before Week 25 were deemed to have experienced a BTH event. Percentages have been rounded off to the first decimal point.
Time Frame: Baseline, Week 25
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Crovalimab
Number analyzed (Participants) | 51
percentage of participants | 3.9 [0.68 to 14.59]

4. Secondary Outcome: Percentage of Participants With Stabilized Hemoglobin
Description: Stabilized hemoglobin was defined as avoidance of a ≥2 g/dL decrease in hemoglobin level from baseline, in the absence of transfusion. As pre-specified in the SAP participants withdrawing before Week 25 were deemed to not have hemoglobin stabilization.
Time Frame: Baseline, Week 25
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Crovalimab
Number analyzed (Participants) | 51
percentage of participants | 51.0 [36.77 to 65.05]

5. Secondary Outcome: Change From Baseline in Fatigue in Adults Aged >=18 Years
Description: Fatigue was assessed using functional assessment of chronic illness therapy-fatigue (FACIT-F) scale. FACIT-F is a self-assessment questionnaire with a 7-day recall period and 13 items evaluating fatigue and its impact on daily life activities. Items are scored on a response scale that ranges from 0 ("not at all") to 4 ("very much so"). Relevant items are reverse scored, and all the items are summed to create a total score range from 0 to 52, with 0 being the worst possible score and 52 being the best possible score. A higher score indicates low fatigue severity. A positive mean change indicates improvement. FACIT-F was assessed in adult participants only. FACIT-F assessment was unintentionally missed in the Schedule of Activities (SoA) table, which site used to guide the assessments at each timepoint. Therefore, data were not collected at Week 25.
Time Frame: Baseline, Week 2, Week 5, Week 9, Week 17, Week 25
Population: PAP included all enrolled participants who received at least one dose of crovalimab and had at least one central LDH level assessment after the first IV infusion. Overall number analyzed is the number of participants ≥18 years with data available for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crovalimab
Number analyzed (Participants) | 48
score on a scale
  Baseline | 31.77 (8.53)
  Change from Baseline at Week 2 | 6.67 (8.02)
  Change from Baseline at Week 5 | 8.08 (9.28)
  Change from Baseline at Week 9 | 8.15 (10.61)
  Change from Baseline at Week 17 | 8.77 (9.63)
  Change from Baseline at Week 25: number analyzed (Participants) | 0

6. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Time Frame: Up to 7 years
Reporting Status: Not Posted, anticipated posting 2029-02

7. Secondary Outcome: Percentage of Participants With Injection-Site Reactions, Infusion-Related Reactions, Hypersensitivity, and Infections (Including Meningococcal Meningitis)
Time Frame: Up to 7 years
Reporting Status: Not Posted, anticipated posting 2029-02

8. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) Leading to Study Drug Discontinuation
Time Frame: Up to 7 years
Reporting Status: Not Posted, anticipated posting 2029-02

9. Secondary Outcome: Trough Serum Concentration of Crovalimab Over Time
Time Frame: Up to 7 years
Reporting Status: Not Posted, anticipated posting 2029-02

10. Secondary Outcome: Serum Concentrations of Crovalimab
Time Frame: Up to 7 years
Reporting Status: Not Posted, anticipated posting 2029-02

11. Secondary Outcome: Percentage of Participants With Anti-Drug Antibodies (ADAs) to Crovalimab
Time Frame: Up to 7 years
Reporting Status: Not Posted, anticipated posting 2029-02

12. Secondary Outcome: Terminal Complement Activity as Measured by Liposome Immunoassay (LIA)
Time Frame: Up to 7 years
Reporting Status: Not Posted, anticipated posting 2029-02

13. Secondary Outcome: Change Over Time in Total and Free C5 Concentration
Time Frame: Up to 7 years
Reporting Status: Not Posted, anticipated posting 2029-02

14. Secondary Outcome: Observed Value in Absolute Reticulocyte Count
Time Frame: Up to 7 years
Reporting Status: Not Posted, anticipated posting 2029-02

15. Secondary Outcome: Observed Value in Free Hemoglobin
Time Frame: Up to 7 years
Reporting Status: Not Posted, anticipated posting 2029-02

16. Secondary Outcome: Observed Value in Haptoglobin
Time Frame: Up to 7 years
Reporting Status: Not Posted, anticipated posting 2029-02

17. Secondary Outcome: Percent Change From Baseline in Absolute Reticulocyte Count
Time Frame: Baseline, Week 25
Population: Safety population included all enrolled participants who received at least one dose of crovalimab. Number of participants analyzed is the number of participants with data available for analysis at the specified timepoints.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Crovalimab
Number analyzed (Participants) | 44
percent change | 40.9411 (66.0292)

18. Secondary Outcome: Percent Change From Baseline in Free Hemoglobin
Time Frame: Baseline, Week 25
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Crovalimab
Number analyzed (Participants) | 37
percent change | -45.6180 (51.8421)

19. Secondary Outcome: Percent Change From Baseline in Haptoglobin
Time Frame: Baseline, Week 25
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Crovalimab
Number analyzed (Participants) | 37
percent change | 295.1351 (1735.4180)

ADVERSE EVENTS:
Time Frame: From enrollment until primary completion date cutoff (up to approximately 25 weeks)
Description: Safety population included all enrolled participants who received at least one dose of crovalimab.
Arm/Group | CROVALIMAB
All-Cause Mortality (participants affected / at risk) | 1/51
Serious Adverse Events (participants affected / at risk) | 4/51
Other Adverse Events (participants affected / at risk) | 46/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CROVALIMAB (N=51)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Abdominal wall mass (Gastrointestinal disorders) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CROVALIMAB (N=51)
Neutropenia (Blood and lymphatic system disorders) | 7 (8)
Gingival swelling (Gastrointestinal disorders) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 24 (26)
Urinary tract infection (Infections and infestations) | 3 (4)
Alanine aminotransferase increased (Investigations) | 11 (15)
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 8 (8)
Bilirubin conjugated increased (Investigations) | 15 (27)
Blood alkaline phosphatase increased (Investigations) | 9 (12)
Blood bilirubin increased (Investigations) | 9 (10)
Blood bilirubin unconjugated increased (Investigations) | 12 (13)
Gamma-glutamyltransferase increased (Investigations) | 6 (9)
Lymphocyte count decreased (Investigations) | 8 (15)
Neutrophil count decreased (Investigations) | 13 (25)
Platelet count decreased (Investigations) | 5 (10)
Weight increased (Investigations) | 6 (6)
White blood cell count decreased (Investigations) | 12 (29)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 (5)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 5 (16)
Hyperuricaemia (Metabolism and nutrition disorders) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-11-23): https://cdn.clinicaltrials.gov/large-docs/68/NCT04654468/Prot_002.pdf
  • Statistical Analysis Plan (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/68/NCT04654468/SAP_001.pdf